CLINICAL TRIAL: NCT01003561
Title: Hemodynamic Changes of Upper and Lower Extremities After Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Hae K Kil, Severance Hospital, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2009-TURP
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Hypertension
Keywords: ultrasonographic exam on upper and lower extremities
MeSH Terms: conditions — Hypertension | interventions — Anesthesia, Spinal; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Investigator

ARMS (1):
- ultrasonographic exam (Experimental)
  Interventions: Procedure: spinal anesthesia for surgery

INTERVENTIONS:
Procedure: spinal anesthesia for surgery — spinal anesthesia (T10) for elective TURP surgery

SUMMARY:
The aim of this study is to evaluate the changes of venous flow, volume, and resistance in upper (basilic v.) and lower (popliteal v.) extremities of the elderly healthy patients compared with elderly hypertensive patients who undergoing spinal anesthesia for transurethral prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* > 65yr men
* who undergoes spinal anesthesia for elective TURP
* normotensive/hypertensive

Exclusion Criteria:

* vascular disease
* contraindications for spinal anesthesia

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)

PRIMARY OUTCOMES:
Blood flow | during 30 min after spinal anesthesia
Blood volume | during 30 min after spinal anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University, Seoul, South Korea